CLINICAL TRIAL: NCT06368440
Title: A Single-blind, Randomized, Placebo-controlled Study to Investigate the Safety, Tolerability and Pharmacokinetics of an Oral Suspension of AZD6793 Following Single and Multiple Doses in Japanese and Chinese Healthy Participants
Brief Title: A Study to Investigate the Safety and Pharmacokinetics of AZD6793 in Healthy Japanese and Chinese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Other
Other Study IDs: D7860C00003
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Healthy Participants
Keywords: Chronic obstructive pulmonary disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1: Cohort 1 AZD6793 (Experimental): 6 Healthy Japanese participants will receive single dose of AZD6793 dose 1 and 2 healthy Japanese participants will receive matching placebo to AZD6793 as oral suspension on Day 1.
  Interventions: Drug: AZD6793; Drug: Placebo
- Part 1: Cohort 2 AZD6793 (Experimental): 6 Healthy Japanese participants will receive single dose of AZD6793 dose 2 and 2 healthy Japanese participants will receive matching placebo to AZD6793 as oral suspension on Day 1.
  Interventions: Drug: AZD6793; Drug: Placebo
- Part 1: Cohort 3 AZD6793 (Experimental): 6 Healthy Chinese participants will receive single dose of AZD6793 dose 1 and 2 healthy Chinese participants will receive matching placebo to AZD6793 as oral suspension on Day 1.
  Interventions: Drug: AZD6793; Drug: Placebo
- Part 2: Cohort 1 AZD6793 (Experimental): 6 Japanese participants will receive single dose of AZD6793 and 2 participants will receive matching placebo on Day 1. After a washout of at least 48 hours, participants will receive AZD6793 or placebo once daily from Day 3 to Day 8.
  Interventions: Drug: AZD6793; Drug: Placebo
- Part 2: Cohort 2 AZD6793 (Experimental): 6 Chinese participants will receive single dose of AZD6793 and 2 participants will receive matching placebo on Day 1. After a washout of at least 48 hours, participants will receive AZD6793 or placebo once daily from Day 3 to Day 8.
  Interventions: Drug: AZD6793; Drug: Placebo

INTERVENTIONS:
Drug: AZD6793 — Participants will receive AZD6793 single dose as oral suspension.
  Arms: Part 1: Cohort 1 AZD6793; Part 1: Cohort 2 AZD6793; Part 1: Cohort 3 AZD6793
Drug: AZD6793 — Participants will receive AZD6793 multiple doses daily as oral suspension.
  Arms: Part 2: Cohort 1 AZD6793; Part 2: Cohort 2 AZD6793
Drug: Placebo — Participants will receive matching doses of placebo as oral suspension.

SUMMARY:
The main purpose of this study is to assess the safety, tolerability and pharmacokinetics (PK) of oral AZD6793 in healthy Japanese and Chinese participants.

DETAILED DESCRIPTION:
This study will be conducted to assess the safety, tolerability, and PK of oral AZD6793 suspension following single (Part 1) and multiple (Part 2) administrations in healthy Japanese and Chinese participants performed at a single Clinical Unit.

Part 1 of the study will comprise:

* A Screening Period of maximum 28 days (Day -29 to Day -2).
* A Treatment Period during which participants will be resident at the Clinical Unit from Day -1 until at least 72 hours after study intervention administration.
* A Follow-up Visit within 6 ± 1 days after the study intervention administration.

Part 2 of the study will comprise:

* A Screening Period of maximum 28 days (Day -29 to Day -2).
* A Treatment Period during which participants will be resident at the Clinical Unit from Day -1 (the day before first study intervention administration [Day 1]) until Day 10.
* A Follow-up Visit within 6 ± 1 days after the last study intervention administration.

Participants will be randomized to receive AZD6793 and placebo in both Part 1 and Part 2.

Participants who enrolled in Part 1 will be excluded from participation in Part 2 of the study.

ELIGIBILITY:
Main Inclusion Criteria:

1. For Japanese participants only:

   1. Participant was born in Japan
   2. Participant has 2 Japanese biological parents and 4 Japanese grandparents as confirmed by the interview.
   3. Participant did not live outside of Japan for more than 10 years at the time of the Screening Visit.
2. For Chinese participants only:

   1. Participant was born in China (including Hong Kong, Macau, and Taiwan)
   2. Participant has 2 Chinese biological parents and 4 Chinese grandparents as confirmed by the interview.
   3. Participant did not live outside of greater China for more than 10 years at the time of the Screening Visit.
3. All females must have a negative pregnancy test at the Screening Visit and on admission to the Clinical Unit.
4. Females of childbearing potential must not be lactating and if heterosexually active must agree to use an approved method of highly effective contraception,
5. Have a body mass index between 18 and 30 kilograms per meter square (kg/m2) inclusive and weigh at least 45 kilograms (kg), at the Screening Visit.
6. Females of non-childbearing potential must be confirmed at the screening Visit by fulfilling one of the following criteria:

   1. Postmenopausal defined as amenorrhea for at least 12 months following cessation of all exogenous hormonal treatments and FSH levels in the postmenopausal range.
   2. Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy (but not tubal ligation).

Main Exclusion Criteria:

1. History of any clinically important disease or disorder or presence of gastrointestinal, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.

3. Diagnosis or history of immunodeficiency or increased susceptibility to severe infection, or a clinically significant infection within 4 weeks of the Screening Visit.

4. Any positive result on screening for serum hepatitis B surface antigen, hepatitis B core antibody, or human immunodeficiency virus.

5. History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the Investigator or history of hypersensitivity to drugs with a similar chemical structure or class to AZD6793.

6. Plasma donation within one month of the Screening Visit or any blood donation/blood loss greater than (>) 500 milliliter (mL) during the 3 months prior to the Screening Visit.

7. Participants who have previously received AZD6793. 8. Positive or indeterminate QuantiFERON® TB test at Screening Visit. 9. Current smokers or those who have smoked or used nicotine products (including e-cigarettes) within the previous 3 months prior to the Screening Visit.

10. Known or suspected history of alcohol or drug abuse or excessive intake of alcohol as judged by the Investigator.

11. Positive screen for drugs of abuse, or alcohol or cotinine at the Screening Visit or admission to the Clinical Unit (Day -1).

12. Excessive intake of caffeine-containing drinks or food (eg, coffee, tea, chocolate) defined as the regular consumption of more than 500 mg of caffeine per day (eg, > 5 cups of coffee [one cup ~100 mg caffeine]; one cup of tea ~30 mg caffeine).

13. Use of drugs with enzyme inducing properties such as St John's Wort within 3 weeks prior to the first administration of study intervention.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2024-12-23 (Actual)

PRIMARY OUTCOMES:
Part 1 (SAD): Number of Participants with Adverse Events | From Day 1 up to Follow up visit (Day 7±1)
  To assess the safety and tolerability of AZD6793 following oral administration of single ascending doses in healthy Japanese participants and a single dose in healthy Chinese participants.
Part 2 (MAD): Number of Participants with Adverse Events | From Day 1 up to Follow up visit (Day 14±1)
  To assess the safety and tolerability of AZD6793 following oral administration of multiple doses in healthy Japanese and Chinese participants.

SECONDARY OUTCOMES:
Part 1 (SAD) : Maximum Observed Plasma Drug Concentration | Day 1 to Day 3
  To characterize PK of AZD6793 following oral administration of single ascending doses in healthy Japanese participants and a single dose in healthy Chinese participants.
Part 1 (SAD): Time to Reach Peak Concentration (tmax) | Day 1 to Day 3
  To characterize PK of AZD6793 following oral administration of single ascending doses in healthy Japanese participants and a single dose in healthy Chinese participants.
Part 1 (SAD): Terminal Rate Constant, Estimated by Log-Linear Least Squares Regression of the Terminal Part of The Concentration-Time Curve (λz) | Day 1 to Day 3
  To characterize PK of AZD6793 following oral administration of single ascending doses in healthy Japanese participants and a single dose in healthy Chinese participants.
Part 1 (SAD): Half-life Associated with Terminal Slope of a Semi-Logarithmic Concentration-Time Curve (t1/2λz) | Day 1 to Day 3
  To characterize PK of AZD6793 following oral administration of single ascending doses in healthy Japanese participants and a single dose in healthy Chinese participants.
Part 1 (SAD): Partial Area Under the Plasma Concentration Time Curve from Time Zero to Time 12 (AUC[0-12]) | Day 1 to Day 3
  To characterize PK of AZD6793 following oral administration of single ascending doses in healthy Japanese participants and a single dose in healthy Chinese participants.
Part 1 (SAD): Partial Area Under the Plasma Concentration Time Curve from Time Zero to Time 24 (AUC[0-24]) | Day 1 to Day 3
  To characterize PK of AZD6793 following oral administration of single ascending doses in healthy Japanese participants and a single dose in healthy Chinese participants.
Part 1 (SAD): Area Under the Plasma Concentration Curve from Time Zero to the Last Quantifiable Concentration (AUClast) | Day 1 to Day 3
  To characterize PK of AZD6793 following oral administration of single ascending doses in healthy Japanese participants and a single dose in healthy Chinese participants.
Part 1 (SAD): Area Under the Plasma Concentration Time Curve from Time Zero to Infinity (AUCinf) | Day 1 to Day 3
  To characterize PK of AZD6793 following oral administration of single ascending doses in healthy Japanese participants and a single dose in healthy Chinese participants.
Part 1 (SAD): Apparent Total Body Clearance of Drug from Plasma After Extravascular Administration (CL/F) | Day 1 to Day 3
  To characterize PK of AZD6793 following oral administration of single ascending doses in healthy Japanese participants and a single dose in healthy Chinese participants.
Part 1 (SAD): Volume of Distribution (Apparent) at Steady State Following Extravascular Administration (Vz/F) | Day 1 to Day 3
  To characterize PK of AZD6793 following oral administration of single ascending doses in healthy Japanese participants and a single dose in healthy Chinese participants.
Part 1 (SAD): Dose Normalized AUClast | Day 1 to Day 3
  To characterize PK of AZD6793 following oral administration of single ascending doses in healthy Japanese participants and a single dose in healthy Chinese participants.
Part 1 (SAD): Dose Normalized AUCinf | Day 1 to Day 3
  To characterize PK of AZD6793 following oral administration of single ascending doses in healthy Japanese participants and a single dose in healthy Chinese participants.
Part 1 (SAD): Dose Normalized Cmax | Day 1 to Day 3
  To characterize PK of AZD6793 following oral administration of single ascending doses in healthy Japanese participants and a single dose in healthy Chinese participants.
Part 2 (MAD): Maximum Observed Plasma Drug Concentration (Cmax) | Day 1 to Day 10
  To characterize PK of AZD6793 following oral administration of multiple doses in healthy Japanese and Chinese participants.
Part 2 (MAD) : Concentration at the End of The Dosing Interval (Ctrough) | Day 1 to Day 10
  To characterize PK of AZD6793 following oral administration of multiple doses in healthy Japanese and Chinese participants.
Part 2 (MAD): Temporal Change Parameter (TCP) | Day 1 to Day 10
  To characterize PK of AZD6793 following oral administration of multiple doses in healthy Japanese and Chinese participants.
Part 2 (MAD): Time to Reach Peak Concentration (tmax) | Day 1 to Day 10
  To characterize PK of AZD6793 following oral administration of multiple doses in healthy Japanese and Chinese participants.
Part 2 (MAD): Terminal Rate Constant, Estimated by Log-Linear Least Squares Regression of the Terminal Part of The Concentration-Time Curve (λz) | Day 1 to Day 10
  To characterize PK of AZD6793 following oral administration of multiple doses in healthy Japanese and Chinese participants.
Part 2 (MAD): Half-life Associated with Terminal Slope of a Semi-Logarithmic Concentration-Time Curve (t1/2λz) | Day 1 to Day 10
  To characterize PK of AZD6793 following oral administration of multiple doses in healthy Japanese and Chinese participants.
Part 2 (MAD): Partial Area Under the Plasma Concentration Time Curve from Time Zero to Time 24 (AUC[0-24]) | Day 1 to Day 10
  To characterize PK of AZD6793 following oral administration of multiple doses in healthy Japanese and Chinese participants.
Part 2 (MAD): Area Under the Plasma Concentration Curve from Time Zero to the Last Quantifiable Concentration (AUClast) | Day 1 to Day 10
  To characterize PK of AZD6793 following oral administration of multiple doses in healthy Japanese and Chinese participants.
Part 2 (MAD): Area Under the Plasma Concentration Time Curve from Time Zero to Infinity (AUCinf) | Day 1 to Day 10
  To characterize PK of AZD6793 following oral administration of multiple doses in healthy Japanese and Chinese participants.
Part 2 (MAD): Area Under Plasma Concentration-Time Curve in The Dosing Interval Tau (AUCtau) | Day 1 to Day 10
  To characterize PK of AZD6793 following oral administration of multiple doses in healthy Japanese and Chinese participants.
Part 2 (MAD): Apparent Total Body Clearance of Drug from Plasma After Extravascular Administration (CL/F) | Day 1 to Day 10
  To characterize PK of AZD6793 following oral administration of multiple doses in healthy Japanese and Chinese participants.
Part 2 (MAD): Volume of Distribution (Apparent) at Steady State Following Extravascular Administration (Vz/F) | Day 1 to Day 10
  To characterize PK of AZD6793 following oral administration of multiple doses in healthy Japanese and Chinese participants.
Part 2 (MAD): Dose Normalized AUClast | Day 1 to Day 10
  To characterize PK of AZD6793 following oral administration of multiple doses in healthy Japanese and Chinese participants.
Part 2 (MAD): Dose Normalized AUCtau | Day 1 to Day 10
  To characterize PK of AZD6793 following oral administration of multiple doses in healthy Japanese and Chinese participants.
Part 2 (MAD): Dose Normalized Cmax | Day 1 to Day 10
  To characterize PK of AZD6793 following oral administration of multiple doses in healthy Japanese and Chinese participants.
Part 2 (MAD): Ratio of the Area Under the Curve (Rac AUC) | Day 1 to Day 10
  To characterize PK of AZD6793 following oral administration of multiple doses in healthy Japanese and Chinese participants.
Part 2 (MAD): Accumulation Ratio Based on Cmax (Rac Cmax) | Day 1 to Day 10
  To characterize PK of AZD6793 following oral administration of multiple doses in healthy Japanese and Chinese participants.
Part 2 (MAD): Amount of Unchanged Drug Excreted into Urine from Time t1 to Time t2 (Ae[t1-t2]) | Days 1, 2, and 8
  To characterize PK of AZD6793 in urine following oral administration of multiple doses in healthy Japanese and Chinese participants.
Part 2 (MAD): Cumulative Amount of Unchanged Drug Excreted into Urine (Aeinf) | Days 1, 2, and 8
  To characterize PK of AZD6793 in urine following oral administration of multiple doses in healthy Japanese and Chinese participants.
Part 2 (MAD): Renal Clearance (CLR) | Days 1, 2, and 8
  To characterize PK of AZD6793 in urine following oral administration of multiple doses in healthy Japanese and Chinese participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure."Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure researchenvironmentVivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- See also: D7860C00003_CSR Synopsis_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D7860C00003&attachmentIdentifier=136fad38-bc6c-48b3-a26a-021b8f22a5e9&fileName=D7860C00003_CSR_Synopsis_Redacted.pdf&versionIdentifier=